CLINICAL TRIAL: NCT06013605
Title: Effect of Walking Exercise on Functional Capacity and Productivity in Patients After Coronary Artery Bypass Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Indra Gilang Pamungkas, Ns. Indra Gilang Pamungkas, S.Kep., M.Kep, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DP.04.03/KEP064/EC043/2023
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Coronary Artery Bypass; Cardiac Rehabilitation
Keywords: Coronary Artery Bypass; Walking; Functional Capacity; Productivity

STUDY DESIGN:
Intervention Model Description: This study used a parallel Randomized Controlled Trial (RCT) with a 1:1 ratio.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were not involved during the intervention process. Respondents were also asked not to inform the outcome assessor of the measures they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants did walking exercise and usual care (leg straightening)
  Interventions: Behavioral: Walking Exercise and Leg Straightening
- Control Group (Experimental): Participants did usual care (leg straightening)
  Interventions: Behavioral: Leg Straightening

INTERVENTIONS:
Behavioral: Walking Exercise and Leg Straightening — Participants performed the exercise on the day agreed upon with the researcher. Respondents did walking exercises 3 times per week for 4 weeks with a duration of 10 minutes of warm-up, 30 minutes of walking exercises, and 10 minutes of cooling down. Respondents also did leg straightening every day for 4 weeks with a frequency of 1 time a day for 10 minutes.
  Arms: Intervention Group
Behavioral: Leg Straightening — Respondents did leg straightening every day for 4 weeks with a frequency of 1 time a day for 10 minutes.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to assess the effect of walking exercise on functional capacity and productivity in patients after Coronary Artery Bypass Graft who have completed phase II cardiac rehabilitation. The main question it aims to answer are:

1. What is the effect of walking exercise on functional capacity and productivity in patients after Coronary Artery Bypass Graft? Participants performed the exercise on the day agreed upon with the researcher. Respondents did walking exercises 3 times per week for 4 weeks with a duration of 10 minutes of warm-up, 30 minutes of walking exercises, and 10 minutes of cooling down. Respondents also did leg straightening every day for 4 weeks with a frequency of 1 time a day for 10 minutes. Researchers compared between intervention and control group to see if the effect between respondents who did walking and leg straightening exercises and also respondents who only did leg straightening.

DETAILED DESCRIPTION:
The research process was guided by The Consort Statement for RCT research. The process was conducted through the stages of enrollment, allocation, follow-up, and analysis. The recruitment process begins with an eligibility assessment process for potential respondents. This process was carried out when the patient conducted a phase 2 cardiac rehabilitation evaluation. Researchers initially checked patient data through medical records by looking at color codes (pink indicates Coronary Artery Bypass Graft patients), age, and location of residence. The patient's communication skills were observed during the evaluation process. The doctor determines the patient's risk stratification after the evaluation, then the researcher sees the patient's risk stratification from the assessment results in the medical record. The inclusion criteria in this study were patients aged 18-60 years, working, having mild to moderate risk stratification, living in the Jakarta, Bogor, Depok, Tangerang and Bekasi areas, and patients who could communicate well. Respondents who had been collected were then randomized using an envelope so that the respondents were divided into 2 groups where 21 respondents entered the intervention group and 21 respondents entered the control group.

ELIGIBILITY:
Inclusion Criteria:

* Post- CABG patients in phase III of cardiac rehabilitation;
* Patients living in the JaBoDeTaBek area;
* Patients aged 18 - 60 years;
* Patients who have mild to moderate risk stratification;
* Patients who do not have limitations in mobilization such as using mobility aids (wheelchairs, walkers, crutches);
* Patients who do not perform routine aerobic exercise based on time intervals and types of exercise (such as cardiac exercise, cycling, ergocycle, etc.);
* Patients can communicate well and are willing to become respondents by signing informed consent.

Exclusion Criteria:

* Patients with conditions that contraindicate exercise or rehabilitation such as unstable angina pectoris, resting systolic blood pressure >200 mmHg or diastolic >110 mmHg, clinical aortic valve stenosis, acute systemic disease, uncontrolled atrial or ventricular dysrhythmias, uncontrolled sinus tachycardia, uncompensated heart failure, third-degree atrioventricular block without pacing, active pericarditis or myocarditis, pulmonary thromboembolism, depression or ST-segment elevation at rest, Diabetic Mellitus with uncontrolled blood sugar, thyroiditis, hypokalemia, hyperkalemia, hypovolemia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-05-26 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Functional Capacity | 6 minutes
  The ability of post-CABG patients to be able to perform expected activities or workloads can be done using the 6 Minutes Walking Test.
Productivity | 5 minutes
  The ability of post-CABG patients to perform work and physical activities was assessed using the WPAI.

CONTACTS AND LOCATIONS:
Overall Officials: Indra G Pamungkas, Study Chair — Indonesia University
Locations (1):
- National Cardiovascular Center Harapan Kita, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No